CLINICAL TRIAL: NCT07075874
Title: Preoperative Neutrophil-to-Lymphocyte Ratio as a Predictor of Post-Dural Puncture Headache Following Cesarean Section Under Spinal Anesthesia
Brief Title: Neutrophil to Lymphocyte Ratio and Postdural Headache
Status: Recruiting | Type: Observational
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, İlke Dolgun, Assoc. prof, Haseki Training and Research Hospital
Other Study IDs: NLR-PDPH ERKAN
Record Dates: First submitted 2025-07-10; First posted 2025-07-20 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Preoperative Neutrophil-to-Lymphocyte Ratio (NLR); Postdural Puncture Headache
MeSH Terms: conditions — Post-Dural Puncture Headache

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PDPH Group: Patients who developed postdural puncture headache (PDPH) following spinal anesthesia for cesarean section.
  Interventions: Other: PDPH
- Non-PDPH Group: Patients who did not develop PDPH after spinal anesthesia for cesarean section
  Interventions: Other: PDPH

INTERVENTIONS:
Other: PDPH — Observational analysis of preoperative inflammatory markers (e.g., NLR, PLR, SIRI) in relation to PDPH development following spinal anesthesia.

SUMMARY:
This study will aim to investigate whether systemic inflammatory markers-especially the neutrophil-to-lymphocyte ratio (NLR)-obtained from preoperative complete blood counts can predict the development of post-dural puncture headache (PDPH) in obstetric patients undergoing cesarean section under spinal anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 years or older
* Underwent elective or emergency cesarean section under spinal anesthesia
* Had complete preoperative complete blood count (CBC) data available
* No known hematological or inflammatory disease
* No intraoperative complications recorded
* Medical records accessible for postoperative follow-up regarding PDPH symptoms

Exclusion Criteria:

* Age under 18
* Absence of preoperative complete blood count data
* Presence of hematologic malignancy, active infection, autoimmune disease, or immunosuppressive therapy
* Platelet count <150,000/mm³ or INR >1.5
* Incomplete or missing medical records

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only female participants were included, as the study population consisted of obstetric patients undergoing cesarean section under spinal anesthesia.
Study Population: The study population consists of obstetric patients who underwent cesarean section under spinal anesthesia between January 2020 and December 2024 at a single tertiary center.
Sampling Method: Non-Probability Sample
Enrollment: 821 (Estimated)
Dates: Start 2025-07-12 (Actual); Primary Completion 2025-07-15 (Estimated); Study Completion 2025-07-17 (Estimated)

PRIMARY OUTCOMES:
Postdural Puncture Headache (PDPH) incidence | Within 10 days postoperatively
  The occurrence of PDPH symptoms within 10 days following spinal anesthesia in obstetric patients, as documented in medical records.

CONTACTS AND LOCATIONS:
Locations (1):
- Istinye Üniversity, Istanbul, Merkez Mahallesi, Turkey (Türkiye)

REFERENCES:
- [Background] Olawin AM, Das JM. Spinal Anesthesia. 2022 Jun 27. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK537299/ PMID 30725984
- [Result] Sahin R, Tanacan A, Serbetci H, Agaoglu Z, Haksever M, Kara O, Sahin D. The Association of Systemic Immune-Inflammation Index (SII), Systemic Immune-Response Index (SIRI), and Neutrophil-to-Lymphocyte Ratio (NLR) with Cesarean Scar Pregnancy (CSP). J Reprod Immunol. 2024 Aug;164:104275. doi: 10.1016/j.jri.2024.104275. Epub 2024 Jun 4. PMID 38850761
- [Result] Bai YY, Xi Y, Yin BB, Zhang JH, Chen F, Zhu B. Reference intervals of systemic immune-inflammation index, neutrophil-to-lymphocyte ratio, lymphocyte-to-monocyte ratio, and platelet-to-lymphocyte ratio during normal pregnancy in China. Eur Rev Med Pharmacol Sci. 2023 Feb;27(3):1033-1044. doi: 10.26355/eurrev_202302_31199. PMID 36808350